CLINICAL TRIAL: NCT02874404
Title: A Single-Center Phase IIa Study Evaluating the Safety and Tolerability of TGR-1202 and Ibrutinib in Patients With Relapsed or Refractory Diffuse Large B-Cell Lymphoma: A Trial of the Lymphoma Precision Medicine Laboratory
Brief Title: TGR-1202 and Ibrutinib in Treating Patients With Relapsed or Refractory Diffuse Large B-Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0345-16-FB; NCI-2016-01082 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA036727 (NIH)
Record Dates: First submitted 2016-08-17; First posted 2016-08-22 (Estimated); Results first posted 2020-02-26 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: Recurrent Diffuse Large B-Cell Lymphoma; Refractory Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — ibrutinib; umbralisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group A (PI3K delta inhibitor TGR-1202, ibrutinib) (Experimental): Patients receive PI3K delta inhibitor TGR-1202 PO QD on days 1-28 and ibrutinib PO QD on days 9-28 of course 1 and days 1-28 of subsequent courses. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ibrutinib; Other: Laboratory Biomarker Analysis; Drug: PI3K-delta Inhibitor TGR-1202
- Group B (Ibrutinib, PI3K delta inhibitor TGR-1202) (Experimental): Patients receive ibrutinib PO QD on days 1-28 and PI3K delta inhibitor TGR-1202 PO QD and days 9-28 of course 1 and days 1-28 of subsequent courses. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ibrutinib; Other: Laboratory Biomarker Analysis; Drug: PI3K-delta Inhibitor TGR-1202
- Group C (PI3K delta inhibitor TGR-1202, ibrutinib) (Experimental): Patients then receive PI3K delta inhibitor TGR-1202 PO QD and ibrutinib PO QD on days 1-28. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ibrutinib; Other: Laboratory Biomarker Analysis; Drug: PI3K-delta Inhibitor TGR-1202

INTERVENTIONS:
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA-032765; Imbruvica; PCI-32765
Other: Laboratory Biomarker Analysis — Correlative markers
Drug: PI3K-delta Inhibitor TGR-1202 — Given PO
  Other Names: RP5264; TGR-1202

SUMMARY:
This phase IIa trial studies the side effects and how well TGR-1202 and ibrutinib work in treating patients with diffuse large B-cell lymphoma that has returned after a period of improvement or does not respond to treatment. TGR-1202 and ibrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and tolerability of PI3K delta inhibitor TGR-1202 (TGR-1202) and ibrutinib in relapsed and refractory (rel/ref) diffuse large B-cell lymphoma (DLBCL).

SECONDARY OBJECTIVES:

I. To determine the overall response rate (ORR) defined as the sum of complete responses (CR) and partial responses (PR).

II. To determine the event-free survival (EFS), time to response (TTR), and duration of response (DOR) in patients with rel/ref DLBCL.

TERTIARY OBJECTIVES:

I. To evaluate molecular profiling of patient samples (optional lymph node biopsies) obtained at days 0 (pre-treatment; core biopsy), day 8 (fine needle aspiration) and end of treatment (progressive disease or end of study treatment-1 year; core biopsy).

II. To evaluate the baseline characteristics and dynamic shifts in mutational Landscape, transcriptional signatures and intracellular signaling cascades in primary tumor cells.

III. To define the mutational status of 384 genes that mutated in DLBCL, including cluster of differentiation (CD)79B, caspase recruitment domain family member 11 (CARD11), and myeloid differentiation primary response 88 (MYD88).

IV. To evaluate signatures of B-cell receptor signaling and the back-up pathway of oxidative phosphorylation.

V. To measure the basal and induced level of activation of components within parallel signaling pathways downstream of the B-cell receptor.

VI. To monitor changes in T-cell characteristics in response to exposure to TGR-1202 and ibrutinib.

VII. To perform quantitative response evaluation by peripheral blood cell-free deoxyribonucleic acid (DNA) sequencing at enrollment, day 8, 1 month, at every response assessment time point compared to standard radiographic response evaluation by positron emission tomography (PET)/ computed tomography (CT) or CT and end of treatment (progressive disease or end of study treatment-1 year).

VIII. To evaluate the genetic profiling for drug resistance mutations. IX. To evaluate DLBCL subtype analysis by immunohistochemistry compared to Nanostring assessment.

OUTLINE: Patients are assigned to 1 of 3 groups.

GROUP A: Patients receive PI3K delta inhibitor TGR-1202 orally (PO) once daily (QD) on days 1-28 and ibrutinib PO QD on days 9-28 of course 1 and days 1-28 of subsequent courses. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

GROUP B: Patients receive ibrutinib PO QD on days 1-28 and PI3K delta inhibitor TGR-1202 PO QD and days 9-28 of course 1 and days 1-28 of subsequent courses. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

GROUP C: Patients then receive PI3K delta inhibitor TGR-1202 PO QD and ibrutinib PO QD on days 1-28. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days and after 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diffuse large B-cell lymphoma (DLBCL) or transformed DLBCL
* Hematoxylin and eosin (H&E) stain and immunohistochemistry (IHC) slides or a representative formalin-fixed, paraffin-embedded (FFPE) tissue block along with the pathology report from initial diagnosis, (as well as, an optional 8 unstained slides of 4 micron thickness to store for future IHC and DNA specified research use), should be sent to be reviewed, and the diagnosis confirmed by University of Nebraska Medical Center (UNMC) (retrospective diagnostic review: treatment may commence prior to the UNMC review); please NOTE: the diagnostic H&E slide and IHC slides will be returned after review; only the optional 8 unstained slides will be retained and stored for future unspecified research use
* Patients with relapsed or refractory DLBCL that has relapsed post-transplant or that has been determined to be ineligible or unsuitable for transplant; patients must have to have received at least one prior systemic therapy
* Patients must have measurable (>= 1.5 cm) or evaluable disease; baseline measurements and evaluations must be obtained within 6 weeks of registration to the study; abnormal PET scans will not constitute evaluable disease, unless verified by CT scan or other appropriate imaging; measurable disease must have at least one objective measurable disease parameter; a clearly defined, bi-dimensionally measurable defect or mass measuring at least 1.5 cm in diameter on a CT scan will constitute measurable disease; proof of lymphoma in the liver is required by a confirmation biopsy; skin lesions can be used as measurable disease provided bi-dimensional measurements are possible
* Absolute neutrophil count (ANC) >= 1.0 x 10^9/L

  * By automated or manual review, whichever is greatest
* Platelets >= 100 x 10^9/L:

  * Unless due to bone marrow infiltration then eligible if platelets > 50 x 10^9/L)
* Total bilirubin =< 1.5 x upper normal limit if documented hepatic involvement with lymphoma, or =< 5 x upper normal limit if history of Gilbert's disease
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x upper limit of normal (ULN) if no liver involvement or =< 5 x the ULN if documented liver involvement
* Creatinine =< 2.0 mg/dL OR calculated creatinine clearance >= 50 mL/min (as calculated by the Cockcroft-Gault method)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 or expected survival duration of > 2 months
* Ability to swallow and retain oral medication
* Women must not be pregnant or breast-feeding

  * All female patients of child-bearing potential must have a negative serum pregnancy test within 2 weeks prior to treatment to rule out pregnancy
  * Pregnancy testing is not required for post-menopausal or surgically sterilized women
* Male and female patients of reproductive potential must agree to follow accepted birth control measures throughout the study period and for 30 days after the last dose of either study drug for females and 3 months after the last dose of study drug for males
* Patient must be able to adhere to the study visit schedule and other protocol requirements
* Patient must be aware of the neoplastic nature of his/her disease and willingly sign (or their legally-acceptable representatives must sign) an informed consent document indicating that they understand the purpose of and procedures required for the study, including biomarkers, and are willing to participate in the study
* No serious disease or condition that, in the opinion of the investigator, would compromise the patient's ability to participate in the study

Exclusion Criteria:

* Currently receiving cancer therapy (i.e., chemotherapy, radiation therapy, immunotherapy, biologic therapy, hormonal therapy, and surgery and/or tumor embolization) or any investigational drug within 7 days of cycle 1/day 1, 14 days of cycle 1/day 1 for limited palliative radiation, and/or five half-live of an oral therapy

  * Corticosteroid therapy started at least 7 days prior to initiation of treatment (prednisone =< 10 mg daily or equivalent) is allowed as clinically warranted); topical or inhaled corticosteroids are permitted
* Major surgery or a wound that has not fully healed within 4 weeks of enrollment
* History of stroke or intracranial hemorrhage within 6 months prior to enrollment
* Requires anticoagulation with warfarin or equivalent vitamin K antagonists (eg, phenprocoumon)
* Vaccinated with live, attenuated vaccines within 4 weeks of enrollment
* Autologous hematologic stem cell transplant within 3 months of study entry
* Allogeneic hematologic stem cell transplant within 12 months of study entry
* Active graft versus-host disease and must not be on immunosuppression
* Wide field radiotherapy within 28 days of cycle 1/day 1 or active side effects of such therapy
* Active hepatitis B (hepatitis B virus [HBV]) or C (hepatitis C virus [HCV]) infection (negative serology required excluding those with are seropositive due to prior vaccination) and/or known history of human immunodeficiency virus (HIV)
* Primary central nervous system involvement only
* Require treatment with strong cytochrome P450 family 3 subfamily A (CYP3A) inhibitors
* Known history of drug-induced liver injury, alcoholic liver disease, primary biliary cirrhosis, ongoing extra-hepatic obstruction caused by stones, cirrhosis of the liver or portal hypertension
* Any life-threatening illness, severe and/or uncontrolled medical condition, or organ system dysfunction, laboratory abnormality, psychiatric illness or other condition which, in the Investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of ibrutinib capsules, put the study outcomes at undue risk or affect their participation in the study such as

  * Symptomatic, or history of documented congestive heart failure New York Heart Association (NYHA) functional classification III-IV (NYHA)
  * Corrected QT interval using Fridericia's formula (QTcF) > 470 msec (unless related to pacemaker) on echocardiogram (EKG) within 7 days of initiation of treatment
  * Angina not well-controlled by medication
  * Poorly controlled or clinically significant atherosclerotic vascular disease including cerebrovascular accident (CVA), transient ischemic attack (TIA), angioplasty, cardiac or vascular stenting within 6 months prior to enrollment
* Prior malignancies within the past 1 year with exception of adequately treated basal cell, squamous cell skin cancer, or thyroid cancer; carcinoma in situ of the cervix or breast; prostate cancer of Gleason grade 6 or less with stable prostate specific antigen (PSA) levels
* Women who are pregnant or breastfeeding; women who agree to stop breastfeeding would be eligible
* Known hypersensitivity to either study drug (TGR-1202 or ibrutinib)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-10-07 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew A Lunning, DO, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were statified to Arms A, B, or C for correlative sample collection purposes only. Clinical study outcomes are not viewed differently among the groups, so subjects are presented as one arm/group.
Groups:
- All Subjects: Patients receive PI3K delta inhibitor TGR-1202 PO QD and ibrutinib PO QD on days 1-28. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | All Subjects
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Subjects: Patients then receive PI3K delta inhibitor TGR-1202 PO QD and ibrutinib PO QD on days 1-28. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
Arm/Group | All Subjects
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.5 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Participants With Adverse Events
Description: Notable serious or recurrent adverse events (SAEs or AEs) of interest occurring across all cycles regardless of attribution assessed using NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Time Frame: Up to 112 days (course 4)
Measure: Number; unit: percentage of participants
Groups:
- All Subjects: Patients receive PI3K delta inhibitor TGR-1202 PO QD on days 1-28 and ibrutinib PO QD on days 9-28 of course 1 and days 1-28 of subsequent courses. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
Arm/Group | All Subjects
Number analyzed (Participants) | 13
percentage of participants
  G 3-4 elevated AST/ALT | 0
  G 3-4 nausea | 15
  G 3-4 diarrhea | 15

2. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as number of patients achieving a best response of complete response or partial response at any disease assessment time point. Response is based on PET/CT (Deauville 3 or less) or CT alone if CR is achieved by PET/CT. Response criteria, modified from the Lugano response criteria. DLBCL is considered FDG avid.
  Complete response:
  Complete disappearance of all detectable clinical evidence of disease and definitely disease-related symptoms if present before therapy.
  Criteria for Partial Response (PR):
  Regression of measurable disease and no new sites
Time Frame: Up to 4 years
Measure: Count of Participants; unit: Participants
Groups:
- All Patients: Patients receive PI3K delta inhibitor TGR-1202 PO QD on days 1-28 and ibrutinib PO QD on days 9-28 of course 1 and days 1-28 of subsequent courses. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
Arm/Group | All Patients
Number analyzed (Participants) | 13
Participants
  Complete Response | 1
  Partial Response | 3

3. Secondary Outcome: Estimated Progression-free Survival (PFS) at 6 Months
Description: PFS is defined as the time between study registration and documented progression or death if no progression was observed.
Time Frame: Time between study registration and documented progression or death if no progression was observed, assessed up to 4 years (6 Month estimate shown)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Patients
Number analyzed (Participants) | 13
percentage of participants | 8 [0.5 to 29]

ADVERSE EVENTS:
Time Frame: Adverse Event reporting is only for TGR 1202 and Ibrutinib "study medications," until 30 days after last administration of study medication. ( approximately 13 months)
Arm/Group | All Patients
All-Cause Mortality (participants affected / at risk) | 8/13
Serious Adverse Events (participants affected / at risk) | 6/13
Other Adverse Events (participants affected / at risk) | 12/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=13)
hypercalcemia (Metabolism and nutrition disorders) | 2 (2)
abdominal pain (Gastrointestinal disorders) | 1 (1)
anemia (Blood and lymphatic system disorders) | 1 (1)
atrial fibrillation (Cardiac disorders) | 1 (1)
Infections and infestations, Other (Infections and infestations) | 1 (1) — diptheroid contaminant
Infections and infestations, Other (Infections and infestations) | 1 (1) — clostridium difficile colitis
confusion (Psychiatric disorders) | 1 (1)
dehydration (Metabolism and nutrition disorders) | 2 (2)
diarrhea (Metabolism and nutrition disorders) | 1 (1)
edema limbs (General disorders) | 1 (1)
fever (General disorders) | 1 (1)
muscle weakness, general (Musculoskeletal and connective tissue disorders) | 1 (1)
hyponatremia (Metabolism and nutrition disorders) | 1 (1)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other, infected port (Surgical and medical procedures) | 1 (1)
enterocolitis infectious (Infections and infestations) | 1 (1)
nausea (Gastrointestinal disorders) | 2 (2)
pain (General disorders) | 1 (1)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
sepsis (Infections and infestations) | 1 (1)
sinus tachycardia (Cardiac disorders) | 1 (1)
vomiting (Gastrointestinal disorders) | 1 (1)
general disorders, other (General disorders) | 1 (1) — weakness
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=13)
alanine aminotransferase increased (Investigations) | 4 (8)
nausea (Gastrointestinal disorders) | 6 (8)
diarrhea (Gastrointestinal disorders) | 3 (7)
Aspartate aminotransferase increased (Investigations) | 4 (6)
alkaline phosphatase increased (General disorders) | 2 (4)
Fever (General disorders) | 2 (4)
abdominal pain (Gastrointestinal disorders) | 2 (3)
cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
upper respiratory infection (Infections and infestations) | 3 (3)
chills (General disorders) | 2 (2)
Infections and infestations, Other (Infections and infestations) | 1 (2) — clostridium difficile colitis
Other, decreased appetite (Metabolism and nutrition disorders) | 2 (2)
dysphagia (Gastrointestinal disorders) | 2 (2)
headache (Nervous system disorders) | 2 (2)
hyperkalemia (Metabolism and nutrition disorders) | 1 (2)
hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Other, left shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (2)
platelet count decreased (Investigations) | 1 (2)
Other, skin rash (Skin and subcutaneous tissue disorders) | 1 (2)
sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
vomiting (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-07): https://cdn.clinicaltrials.gov/large-docs/04/NCT02874404/Prot_SAP_000.pdf
  • Informed Consent Form (2018-10-25): https://cdn.clinicaltrials.gov/large-docs/04/NCT02874404/ICF_001.pdf